CLINICAL TRIAL: NCT03949166
Title: Does Oral Intake During Labor and Delivery Have an Effect on Complications and Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MMC19-0258-17CTIL
Record Dates: First submitted 2019-05-12; First posted 2019-05-14 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Labor and Delivery
Keywords: labor; delivery; eating
MeSH Terms: interventions — Parturition

STUDY DESIGN:
Intervention Model Description: There are 2 arms - fasting and eating
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting (No Intervention): After completion of an epidural block patients that agreed to participate in the study and were randomised to the fasting arm will be allowed to drink water and clear fluids during labor and delivery as accepted by the institute protocol.
- Eating (Experimental): After completion of an epidural block patients that agreed to participate in the study and were randomized to the eating arm will be allowed to eat during their labor and delivery. They will be provided with the list of food that was approved and accepted by the anesthesia team. They will be asked to try eating every 2 hours but if they feel lack of need to eat or any side effects preventing them to eat they can choose not to eat. When reaching full dilatation of 10cm they will ber asked to stop eating.
  Interventions: Other: food during labor and delivery

INTERVENTIONS:
Other: food during labor and delivery — The food that will be allowed during labor and delivery was approved by the anesthesia team. It includes - fruits, energy bars, yogurt,
  Arms: Eating

SUMMARY:
The recommendations regarding eating and drinking during the labor and delivery process are not clear.

The objective of this study is to assess whether eating and drinking during the labor process improves obstetric outcomes and maternal satisfaction.

Patients admitted for the birthing center during the first stage of the delivery and after having a regional anesthesia are instructed as a routine in our birthing center for fasting and drinking only water and clear fluids during their stay at the labor and delivery room and until after giving birth.

The patients will be asked if they are interested in participating in the study. A patient that is interested will be randomized to join one of the two arms: Fasting arm, with the routine management of water and clear fluids or eating, she will be asked to eat every 2 hours or less a food from a list supplied by the study team.

The list of food was created with the anesthesiologist team according the review board demand.

The data regarding the patients' history, pregnancy and labor and delivery process. Obstetrical and neonatal outcome will be collected. A satisfactory questioner well be sent to all participants.

DETAILED DESCRIPTION:
Vaginal birth can be a prolonged process, especially during the first delivery. The recommendations regarding eating and drinking during the labor and delivery process are not clear. There is no agreement between the physicians regarding eating and drinking while being in labor in the birthing center. This disagreement is due to lack of research in this field and inconclusive results in previous studies.

Prolonged fasting during labor can lead to execution of the patients making them tired and less tolerant to the pain, decreasing their ability to cooperate during the pushing phase. However, the recommendation to avoid eating has justified by the risk for unplanned cesarean section which is done under fasting. In general, cesarean sections are done under regional anesthesia but if there is a need for general anesthesia (due to pain or urgency), there is a risk for aspiration if the patient has not been fasting.

We also know that the stomach is clearing slower in the labor process, therefore some recommend fasting during labor.

In recent years there is a decrease in the use of general anesthesia during cesarean sections and since the incidence of aspiration during cesarean section is rare and due to the demand from the patients for autonomy and controlling their labor process including the option of eating the debate regarding eating during labor and delivery is justified.

In 2009 an ACOG(American College of Obstetricians and Gynecologists ) committee report concluded that there is not enough evidence regarding the link between drinking clear fluids and reflux , vomiting and aspiration during labor.

the objective of this study is to assess whether eating and drinking during the labor process improves obstetric outcomes and maternal satisfaction.

Patients admitted for the birthing center during the first stage of the delivery and after having a regional anesthesia are instructed as a routine in our birthing center for fasting and drinking only water and clear fluids during their stay at the labor and delivery room and until after giving birth.

The patients will be asked if they are interested in participating in the study. A patient that is interested will be randomized to join one of the two arms:

1. Fasting arm- The patient will be allowed to drink water and clear fluids as the routine management in our birthing center
2. Eating arm - The patient will be asked to eat every 2 hours or less a food from a list supplied by the study team, with no limitations on drinking.

The list of food was created with the anesthesiologist team according the review board demand.

The data regarding the patients' history, pregnancy and labor and delivery process. Obstetrical and neonatal outcome will be collected. A satisfactory questioner well be sent to all participants.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy at 37 weeks or more
* After an epidural anaesthesia

Exclusion Criteria:

* Preterm delivery before 37 weeks of pregnancy
* Known anomalies or chromosomal abnormalities
* Patient at increased risk for aspiration based on anesthesiologist assesment
* A patient post epidural anesthesia with pain indicating the need for a new epidural insertion

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-12-18 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
prolonged second stage of labor | the delivery
  The mean time from full dilatation to the delivery of the baby on each group
duration of pushing | the delivery
  The mean time from beginning of pushing with the midwife to the delivery of the baby in each group
operative vaginal delivery | the delivery
  The mean incidence of operative vaginal delivery in each group
cesarean section | the delivery
  The mean incidence of cesarean section in each group

SECONDARY OUTCOMES:
Maternal satisfaction | from 2 days after delivery until 6 months after the delivery , she will be asked once
  The median satisfaction from the delivery of the mother of the delivery process from 1-11

CONTACTS AND LOCATIONS:
Overall Officials: Gil Shechter Maor, MD, Principal Investigator — Meir Medical hospital
Locations (1):
- Meor Medical hospital, Kfar Saba, Israel